CLINICAL TRIAL: NCT03398421
Title: A Single Centre, Open Label, One Sequence, Cross-over Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of Single Inhaled Doses of Nemiralisib in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics (PK) of Nemiralisib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206874
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Results first posted 2019-06-03 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Nemiralisib; Pharmacokinetics; Itraconazole; Drug-drug Interaction; Cross-over
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nemiralisib; Itraconazole

STUDY DESIGN:
Intervention Model Description: Subjects will receive nemiralisib alone on Day 1 in Period 1 and itraconazole from Day 1 to Day 10 followed by nemiralisib on Day 5 in Period 2.
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects receiving nemiralisib and itraconazole (Experimental): Eligible subjects will receive a single dose of 100 micrograms (mcg) nemiralisib on Day 1 in Period 1. Subjects will also receive a single dose of 200 milligrams (mg) itraconazole in the morning from Day 1 to Day 10 and single dose of 100 mcg nemiralisib on Day 5, one hour after the dose of itraconazole in Period 2. There will be a washout of at least 14 days between the administration of nemiralisib in Period 1 and Period 2.
  Interventions: Drug: Nemiralisib; Drug: Itraconazole

INTERVENTIONS:
Drug: Nemiralisib — Nemiralisib will be given as 100 mcg via ELLIPTA Dry Powder Inhaler with 30 doses per inhaler/ 100 mcg total dose. ELLIPTA® is a registered trademark of GlaxoSmithKline group of companies.
Drug: Itraconazole — Itraconazole will be given as 100 mg per capsule per day administered orally with water

SUMMARY:
Nemiralisib is a potent anti-inflammatory agent for the treatment of chronic obstructive pulmonary disease (COPD) and other inflammatory lung diseases. The Cytochrome P450 3A4 (CYP3A4) is a major route of clearance for nemiralisib. The co-administration of drug therapies, which modulate CYP3A4, may alter the exposure of nemiralisib. Hence, this clinical drug interaction study with itraconazole (a potent CYP3A4 inhibitor) is required. The study will evaluate the PK, safety and tolerability of nemiralisib when administered alone and when administered concomitantly with repeat doses of itraconazole in healthy males and females. Subjects will receive treatment with nemiralisib alone in Period 1 and itraconazole followed by nemiralisib in Period 2 in single sequence crossover manner. Approximately 20 subjects will be enrolled such that approximately 16 evaluable subjects complete the study. Each subject will participate in the study for approximately 7 weeks including screening visit, 2 treatment periods and a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac evaluation.
* Normal spirometry at Screening (FEV1 and forced vital capacity [FVC] >=80 percent of predicted. Measurements to be taken in triplicate. The highest value of each individual component must be >=80 percent of predicted).
* A subject with a clinical abnormality or laboratory parameter(s) (except for liver function tests) outside the reference range for the population being studied may be included only if the investigator, in consultation with the medical monitor if needed, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >50 kilograms (kg) and body mass index (BMI) within the range 18.0-35.0 kg per meter square (kg/m^2) (inclusive).
* Male and/or female: A male subject must agree to use contraception during the treatment period and for at least 10 days after the last dose of study treatment and refrain from donating sperm during this period; a female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory (except childhood asthma, which has now remitted), hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure.
* Liver function test results above the upper limit of normal (ULN).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 90 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Positive human immunodeficiency virus (HIV) antibody test (according to local policies).
* Positive drug/alcohol test at screening or on admission (Day -1).
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 6 months of screening, or a total pack year history of >5 pack years. [number of pack years = (number of cigarettes per day/20) x number of years smoked].
* Sensitivity to any of the study treatments, or components thereof (including lactose and Magnesium Stearate), or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Unwillingness to follow the lifestyle restrictions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20330

REFERENCES:
- [Background] Patel A, Wilson R, Harrell AW, Taskar KS, Taylor M, Tracey H, Riddell K, Georgiou A, Cahn AP, Marotti M, Hessel EM. Drug Interactions for Low-Dose Inhaled Nemiralisib: A Case Study Integrating Modeling, In Vitro, and Clinical Investigations. Drug Metab Dispos. 2020 Apr;48(4):307-316. doi: 10.1124/dmd.119.089003. Epub 2020 Feb 2. PMID 32009006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase I, single center, open label, one sequence cross-over study conducted in healthy males and females of non-child bearing potential to evaluate the pharmacokinetic (PK), safety and tolerability of nemiralisib administered alone and concomitantly with repeated doses of itraconazole.
Pre-assignment Details: A total of 20 participants were enrolled at a single center in the United States.
Groups:
- Nemiralisib 100 mcg: Participants received a single inhaled oral dose of 100 microgram (mcg) nemiralisib on Day 1 of Period 1 followed by a washout period of 14 days.
- Itraconazole 200 Milligram(mg) With 100mcg Nemiralisib: After a washout period of 14 days, participants received a single oral dose of 200 mg Itraconazole from Days 1 to 10. On Day 5, they received a single inhaled oral dose of 100 mcg nemiralisib one hour after the dose of 200 mg Itraconazole.
Period: Treatment Period 1 (Up to 6 Days)
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 Milligram(mg) With 100mcg Nemiralisib
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0
Period: Washout Period (Up to 14 Days)
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 Milligram(mg) With 100mcg Nemiralisib
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0
Period: Treatment Period 2 (Up to 11 Days)
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 Milligram(mg) With 100mcg Nemiralisib
Started | 0 | 20
Completed | 0 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants received a single 100 mcg inhaled oral dose of Nemiralisib on Day 1 in Period 1, followed by a washout period of 14 days. In treatment period 2, participants received an oral dose of 200 mg itraconazole from Days 1 to 10 and on Day 5 a single inhaled oral dose of 100 mcg nemiralisib was administered one hour after itraconazole dosing.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  American Indian or Alaska Native | 1
  Black or African American | 5
  White/ Caucasian/ European Heritage | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of Nemiralisib in Plasma
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate pharmacokinetic parameters of nemiralisib in both treatment period 1 and 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Pharmacokinetic population comprised of all participants enrolled in the study who took at least 1 dose of nemiralisib and for whom a nemiralisib pharmacokinetic sample was obtained and analyzed.
Time Frame: Period 1: Pre-dose, and 5, 30 minutes, 2, 6, 12, 24, 48, 72, 96 and 120 hours post-dose on Day 1. Period 2: Pre-dose, and 5 min, 30 min, 2, 6, 12, 24, 48, 72, 96, 120 and 144 hours post-dose on Day 5
Population: Pharmacokinetic population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Groups:
- Itraconazole 200 mg and 100mcg Nemiralisib on Day 5: After a washout period of 14 days, participants received a single oral dose of 200 mg Itraconazole from Days 1 to 10. On Day 5, they received a single inhaled oral dose of 100 mcg nemiralisib one hour after the dose of 200 mg Itraconazole.
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Hours*picogram per milliliter
  Day 1, n=20, 0: number analyzed (Participants) | 20 | 0
  Day 1, n=20, 0 | 3199.0 (29.8) |
  Day 5, n=0, 14: number analyzed (Participants) | 0 | 14
  Day 5, n=0, 14 |  | 6272.7 (27.5)
Statistical Analysis 1: Comparison: Nemiralisib 100 mcg vs Itraconazole 200 mg and 100mcg Nemiralisib on Day 5; Test type: Superiority; Ratio of adjusted geometric mean = 2.005, 90% CI 2-sided [1.807 to 2.224]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC [0-t]) of Nemiralisib in Plasma
Description: Blood samples were collected from participants at indicated time frames after the administration of study treatment to investigate pharmacokinetic parameters of Nemiralisib in both treatment period 1 and 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Hour*picogram per milliliter
  Day 1; n=20, 0: number analyzed (Participants) | 20 | 0
  Day 1; n=20, 0 | 2677.1 (30.2) |
  Day 5; n=0, 20: number analyzed (Participants) | 0 | 20
  Day 5; n=0, 20 |  | 4802.3 (29.1)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Nemiralisib in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Picogram per milliliter
  Day 1; n=20, 0: number analyzed (Participants) | 20 | 0
  Day 1; n=20, 0 | 478.7 (41.9) |
  Day 5; n=0, 20: number analyzed (Participants) | 0 | 20
  Day 5; n=0, 20 |  | 384.0 (34.0)

4. Primary Outcome: Apparent Terminal Half-life (t1/2) of Nemiralisib in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Hours
  Day 1, n=20, 0: number analyzed (Participants) | 20 | 0
  Day 1, n=20, 0 | 40.03 (21.7) |
  Day 5, n=0, 14: number analyzed (Participants) | 0 | 14
  Day 5, n=0, 14 |  | 64.00 (11.4)

5. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Nemiralisib in Plasma
Description: Blood samples were collected at indicated time points after administration of repeated doses of itraconazole along with Nemiralisib. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Hour
  Day 1; n=20, 0: number analyzed (Participants) | 20 | 0
  Day 1; n=20, 0 | 0.070 [0.07 to 0.08] |
  Day 5; n=0, 20: number analyzed (Participants) | 0 | 20
  Day 5; n=0, 20 |  | 0.088 [0.08 to 0.10]

6. Secondary Outcome: AUC(0-inf) of Itraconazole and Hydroxy Itraconazole When Co-administered With Nemiralisib in Treatment Period 2
Description: as for outcome 5
Time Frame: Pre-dose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post-dose (itraconazole) on Day 1; Pre-dose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose (itraconazole) on Day 5
Population: Pharmacokinetic population. Only those participants with data available at specified time points were analyzed. NA indicates AUC (0-inf) for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Groups:
- Nemiralisib 100 mcg With Itraconazole 200 mg: After a washout period of 14 days, participants received a single oral dose of 200 mg Itraconazole from Days 1 to 10. On Day 5, they received a single inhaled oral dose of 100 mcg nemiralisib one hour after the dose of 200 mg Itraconazole.
Arm/Group | Nemiralisib 100 mcg With Itraconazole 200 mg
Number analyzed (Participants) | 20
Hour*nanogram per milliliter
  Itraconazole, Day 1: number analyzed (Participants) | 7
  Itraconazole, Day 1 | 1201.3 (46.3)
  Itraconazole, Day 5: number analyzed (Participants) | 7
  Itraconazole, Day 5 | NA (NA) — NA indicates AUC (0-inf) for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
  Hydroxy Itraconazole, Day 1: number analyzed (Participants) | 7
  Hydroxy Itraconazole, Day 1 | NA (NA) — NA indicates AUC (0-inf) for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
  Hydroxy Itraconazole, Day 5 | NA (NA) — NA indicates AUC (0-inf) for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.

7. Secondary Outcome: AUC(0-t) of Itraconazole and Hydroxy Itraconazole When Co-administered With Nemiralisib in Treatment Period 2
Description: as for outcome 5
Time Frame: as for outcome 6
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Hour*nanogram per milliliter
  Itraconazole, Day 1 | 891.7 (60.0)
  Itraconazole, Day 5 | 4939.6 (60.2)
  Hydroxy Itraconazole, Day 1 | 1862.6 (48.8)
  Hydroxy Itraconazole, Day 5 | 10106.4 (50.3)

8. Secondary Outcome: Cmax of Itraconazole and Hydroxy Itraconazole When Co-administered With Nemiralisib in Treatment Period 2
Description: Blood samples were collected at indicated time points after administration of repeated doses of Itraconazole and Hydroxy Itraconazole along with Nemiralisib. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 6
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Nanogram per milliliter
  Itraconazole, Day 1 | 156.90 (59.0)
  Itraconazole, Day 5 | 472.52 (63.7)
  Hydroxy Itraconazole, Day 1 | 240.3 (45.2)
  Hydroxy Itraconazole, Day 5 | 541.2 (41.8)
Statistical Analysis 1: Comparison: Itraconazole 200 mg and 100mcg Nemiralisib on Day 5; Test type: Superiority; Ratio of adjusted geometric mean = 0.802, 90% CI 2-sided [0.690 to 0.933]

9. Secondary Outcome: T1/2 of Itraconazole and Hydroxy Itraconazole When Co-administered With Nemiralisib in Treatment Period 2
Description: as for outcome 8
Time Frame: as for outcome 6
Population: Pharmacokinetic population. Only those participants with data available at specified time points were analyzed. NA indicates T1/2 for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 7
Hour
  Itraconazole, Day 1 | 3.865 (7.7)
  Itraconazole, Day 5 | NA (NA) — NA indicates T1/2 for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
  Hydroxy Itraconazole, Day 1 | NA (NA) — NA indicates T1/2 for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.
  Hydroxy Itraconazole, Day 5 | NA (NA) — NA indicates T1/2 for hydroxy itraconazole (Day 1 and Day 5) and Itraconazole (Day 5) could not be calculated as it was not possible to get accurate measurements since the length was too long for sampling.

10. Secondary Outcome: Tmax of Itraconazole and Hydroxy Itraconazole When Co-administered With Nemiralisib in Treatment Period 2
Description: as for outcome 8
Time Frame: as for outcome 6
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Hour
  Itraconazole, Day 1 | 4.001 [2.00 to 6.00]
  Itraconazole, Day 5 | 4.001 [2.00 to 6.00]
  Hydroxy Itraconazole, Day 1 | 4.004 [3.00 to 6.01]
  Hydroxy Itraconazole, Day 5 | 4.004 [3.00 to 8.01]

11. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per Medical or scientific judgement. Safety population comprised of all participants enrolled in the study, who took at least one dose of study treatment.
Time Frame: Up to 35 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Participants
  Any AE | 1 | 4
  Any SAE | 0 | 0

12. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered: Calcium, Glucose, Potassium and Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters including calcium, glucose, potassium and sodium. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Millimoles/Liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Millimoles/Liter
  Glucose | -0.12 (0.247)
  Calcium | 0.06 (0.070)
  Potassium | 0.20 (0.290)
  Sodium | -0.9 (2.05)

13. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Nemiralisib 100 mcg When Co-administered With Itraconazole 200 mg Repeated Dose: Calcium, Glucose, Potassium and Sodium
Description: as for outcome 12
Time Frame: Baseline (Day -1), Day 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Millimoles/Liter
Arm/Group | Nemiralisib 100 mcg With Itraconazole 200 mg
Number analyzed (Participants) | 20
Millimoles/Liter
  Glucose, Day 2 | -0.08 (0.256)
  Glucose, Day 4 | -0.12 (0.291)
  Glucose, Day 6 | 1.22 (1.055)
  Glucose, Day 8 | -0.22 (0.346)
  Glucose, Day 10 | -0.22 (0.280)
  Calcium, Day 2 | 0.02 (0.066)
  Calcium, Day 4 | 0.03 (0.069)
  Calcium, Day 6 | 0.05 (0.081)
  Calcium, Day 8 | 0.00 (0.077)
  Calcium, Day 10 | 0.03 (0.059)
  Potassium, Day 2 | 0.07 (0.326)
  Potassium, Day 4 | 0.29 (0.381)
  Potassium, Day 6 | 0.01 (0.348)
  Potassium, Day 8 | 0.21 (0.323)
  Potassium, Day 10 | 0.20 (0.339)
  Sodium, Day 2 | -1.0 (1.59)
  Sodium, Day 4 | 0.0 (2.55)
  Sodium, Day 6 | -1.6 (1.73)
  Sodium, Day 8 | -1.0 (1.72)
  Sodium, Day 10 | -1.6 (2.09)

14. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered: Alkaline Phosphate, Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including alkaline phosphate, ALT and AST at indicated time points. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: International Units/ Liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
International Units/ Liter
  Alkaline phosphate | 0.8 (8.08)
  ALT | 1.5 (7.40)
  AST | -0.5 (3.40)

15. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Nemiralisib 100 mcg When Co-administered With Itraconazole 200 mg Repeated Dose: Alkaline Phosphate, ALT and AST
Description: as for outcome 14
Time Frame: Baseline, Day 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: International Units/ Liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
International Units/ Liter
  Alkaline phosphate, Day 2 | -7.0 (6.99)
  Alkaline phosphate, Day 4 | -8.5 (7.00)
  Alkaline phosphate, Day 6 | -7.2 (9.09)
  Alkaline phosphate, Day 8 | -7.6 (8.02)
  Alkaline phosphate, Day 10 | -5.3 (9.35)
  ALT, Day 2 | -3.2 (4.46)
  ALT, Day 4 | -3.2 (3.82)
  ALT, Day 6 | -2.9 (3.11)
  ALT, Day 8 | -2.6 (2.96)
  ALT, Day 10 | -2.8 (4.79)
  AST, Day 2 | -2.6 (3.82)
  AST, Day 4 | -3.0 (3.18)
  AST, Day 6 | -2.4 (2.96)
  AST, Day 8 | -3.2 (2.91)
  AST, Day 10 | -2.0 (3.87)

16. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered:Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, direct bilirubin and creatinine at indicated time points. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Micromoles per liter
  Bilirubin | 5.557 (7.2310)
  Direct bilirubin | 2.394 (0.8595)
  Creatinine | -3.094 (6.5872)

17. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters When Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose: Bilirubin, Direct Bilirubin and Creatinine
Description: as for outcome 16
Time Frame: Baseline, Day 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Micromoles per liter
  Bilirubin, Day 2 | 0.428 (2.7670)
  Bilirubin, Day 4 | 1.796 (2.5710)
  Bilirubin, Day 6 | 2.907 (2.9928)
  Bilirubin, Day 8 | 2.309 (2.6766)
  Bilirubin, Day 10 | 3.506 (2.7447)
  Direct bilirubin, Day 2 | 2.907 (0.9768)
  Direct bilirubin, Day 4 | 2.394 (1.0230)
  Direct bilirubin, Day 6 | 1.796 (0.8728)
  Direct bilirubin, Day 8 | 2.052 (0.7018)
  Direct bilirubin, Day 10 | 2.907 (1.3702)
  Creatinine, Day 2 | 0.442 (8.8284)
  Creatinine, Day 4 | 2.210 (7.5202)
  Creatinine, Day 6 | 0.884 (7.5338)
  Creatinine, Day 8 | 0.442 (7.8414)
  Creatinine, Day 10 | 0.000 (8.6042)

18. Secondary Outcome: Change From Baseline of Total Protein When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of total protein at indicated time points. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Gram per liter | 3.3 (3.85)

19. Secondary Outcome: Change From Baseline of Total Protein When Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose
Description: as for outcome 18
Time Frame: Baseline, Day 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Gram per liter
  Day 2 | -3.8 (3.52)
  Day 4 | -3.4 (3.03)
  Day 6 | 0.2 (3.74)
  Day 8 | -2.4 (3.86)
  Day 10 | -1.8 (2.95)

20. Secondary Outcome: Change From Baseline in Hematology Parameters When Single Oral Dose of Nemiralisib 100 mcg Administered: Lymphocytes, Neutrophils, Platelets, Basophils, Eosinophils, Monocytes, Erythrocytes and White Blood Cells (WBC)
Description: Blood samples were collected for the analysis of hematology parameters including lymphocytes, neutrophils, platelets, basophils, eosinophils, monocytes, erythrocytes and WBCs at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
10^9 cells per liter
  Lymphocytes | -0.264 (0.579)
  Neutrophils | 0.198 (0.736)
  Platelets | 8.4 (31.74)
  Basophils | 0.003 (0.014)
  Eosinophils | -0.038 (0.047)
  Monocytes | -0.054 (0.108)
  Erythrocytes | 242.0 (205.16)
  WBC | -0.174 (0.981)

21. Secondary Outcome: Change From Baseline in Hematology Parameters When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose: Lymphocytes, Neutrophils, Platelets, Basophils, Eosinophils, Monocytes, Erythrocytes and WBC
Description: as for outcome 20
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
10^9 cells per liter
  Lymphocytes | -0.202 (0.339)
  Neutrophils | -0.127 (0.659)
  Platelets | -5.7 (28.24)
  Basophils | -0.004 (0.012)
  Eosinophils | 0.003 (0.057)
  Monocytes | -0.014 (0.130)
  Erythrocytes | 76.0 (165.83)
  WBC | -0.366 (0.846)

22. Secondary Outcome: Change From Baseline in Hematocrit When Single Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of hematocrit at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Percentage of red blood cells in blood | 1.94 (2.067)

23. Secondary Outcome: Change From Baseline in Hematocrit When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg
Description: as for outcome 22
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Percentage of red blood cells in blood | 0.14 (1.436)

24. Secondary Outcome: Change From Baseline in Hemoglobin When Single Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of hemoglobin at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Grams per liter | 7.3 (6.00)

25. Secondary Outcome: Change From Baseline in Hemoglobin When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg
Description: as for outcome 24
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Grams per liter | 1.9 (4.42)

26. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin (MCH) When Single Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of MCH at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Picograms per liter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Picograms per liter | -0.03 (0.459)

27. Secondary Outcome: Change From Baseline in MCH When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg
Description: as for outcome 26
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Picograms per liter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Picograms per liter | -0.12 (0.387)

28. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume (MCV) When Single Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of MCV at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Femtoliter | -0.47 (0.889)

29. Secondary Outcome: Change From Baseline in MCV When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg
Description: as for outcome 28
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Femtoliter | -1.09 (0.972)

30. Secondary Outcome: Change From Baseline in Reticulocyte Percentage When Single Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood samples were collected for the analysis of reticulocyte percentage at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Percentage | -0.038 (0.302)

31. Secondary Outcome: Change From Baseline in Reticulocyte Percentage When Single Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg
Description: as for outcome 30
Time Frame: Baseline and Day 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Percentage | 0.065 (0.267)

32. Secondary Outcome: Specific Gravity at Indicated Time Points
Description: Urine samples were collected for analysis of specific gravity of urine. Urinary specific gravity is the measure of the concentration solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine.
Time Frame: Days -1, 6 and 10
Population: Safety population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Grams per cubic centimeter
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Grams per cubic centimeter
  Day -1, n=20, 19: number analyzed (Participants) | 20 | 19
  Day -1, n=20, 19 | 1.0198 (0.00713) | 1.0207 (0.00863)
  Day 6, n=20, 0: number analyzed (Participants) | 20 | 0
  Day 6, n=20, 0 | 1.0188 (0.00614) |
  Day 10, n=0, 20: number analyzed (Participants) | 0 | 20
  Day 10, n=0, 20 |  | 1.0175 (0.00583)

33. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameter
Description: The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters can be read as Trace and 2+ indicating proportional concentrations in the urine sample. Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Days -1, 6 and 10
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Participants
  Ketones, Day -1, Trace, n=20,19: number analyzed (Participants) | 20 | 19
  Ketones, Day -1, Trace, n=20,19 | 2 | 2
  Protein, Day -1, Trace, n=20,19: number analyzed (Participants) | 20 | 19
  Protein, Day -1, Trace, n=20,19 | 0 | 1
  Erythrocytes, Day-1,Trace, n=20,19: number analyzed (Participants) | 20 | 19
  Erythrocytes, Day-1,Trace, n=20,19 | 1 | 0
  Erythrocytes, Day-1,2+, n=20,19: number analyzed (Participants) | 20 | 19
  Erythrocytes, Day-1,2+, n=20,19 | 1 | 1
  Leukocytes, Day 6, Trace, n=20,0: number analyzed (Participants) | 20 | 0
  Leukocytes, Day 6, Trace, n=20,0 | 2 |
  Leukocytes, Day 6, 2+, n=20,0: number analyzed (Participants) | 20 | 0
  Leukocytes, Day 6, 2+, n=20,0 | 1 |

34. Secondary Outcome: Number of Participants With Urine Potential of Hydrogen (pH) at Indicated Time Points
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0).
Time Frame: Day -1, 6 and 10
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Participants
  Day -1, pH=5, n=20,19: number analyzed (Participants) | 20 | 19
  Day -1, pH=5, n=20,19 | 8 | 8
  Day -1, pH=6, n=20,19: number analyzed (Participants) | 20 | 19
  Day -1, pH=6, n=20,19 | 9 | 8
  Day -1, pH=7, n=20,19: number analyzed (Participants) | 20 | 19
  Day -1, pH=7, n=20,19 | 2 | 3
  Day -1, pH=8, n=20,19: number analyzed (Participants) | 20 | 19
  Day -1, pH=8, n=20,19 | 1 | 0
  Day 6, pH=5, n=20,0: number analyzed (Participants) | 20 | 0
  Day 6, pH=5, n=20,0 | 9 |
  Day 6, pH=6, n=20,0: number analyzed (Participants) | 20 | 0
  Day 6, pH=6, n=20,0 | 8 |
  Day 6, pH=7, n=20,0: number analyzed (Participants) | 20 | 0
  Day 6, pH=7, n=20,0 | 3 |
  Day 10, pH=5, n=0,20: number analyzed (Participants) | 0 | 20
  Day 10, pH=5, n=0,20 |  | 9
  Day 10, pH=6, n=0,20: number analyzed (Participants) | 0 | 20
  Day 10, pH=6, n=0,20 |  | 4
  Day 10, pH=7, n=0,20: number analyzed (Participants) | 0 | 20
  Day 10, pH=7, n=0,20 |  | 7

35. Secondary Outcome: Number of Participants With Abnormal Microscopic Examinations: Casts, Epithelial Cells, Erythrocytes and Leukocytes
Description: A microscopic examination was performed as part of a routine urinalysis. The microscopic exam was performed on urine sediment - urine was centrifuged to concentrate the substances in it at the bottom of a tube. The fluid at the top of the tube was then discarded and the drops of fluid remaining were examined under a microscope. Cells, crystals, and other substances were counted and reported either as the number observed "per low power field" (LPF) or "per high power field" (HPF).
Time Frame: Day -1
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Participants
  Cast0, n=2,2: number analyzed (Participants) | 2 | 2
  Cast0, n=2,2 | 1 | 0
  Cast2, n=2,2: number analyzed (Participants) | 2 | 2
  Cast2, n=2,2 | 0 | 1
  Cast3, n=2,2: number analyzed (Participants) | 2 | 2
  Cast3, n=2,2 | 1 | 0
  Cast10, n=2,2: number analyzed (Participants) | 2 | 2
  Cast10, n=2,2 | 0 | 1
  Epithelial cells 0, n=2,2: number analyzed (Participants) | 2 | 2
  Epithelial cells 0, n=2,2 | 2 | 1
  Epithelial cells 1, n=2,2: number analyzed (Participants) | 2 | 2
  Epithelial cells 1, n=2,2 | 0 | 1
  Erythrocytes 1, n=2,2: number analyzed (Participants) | 2 | 2
  Erythrocytes 1, n=2,2 | 1 | 0
  Erythrocytes 3, n=2,2: number analyzed (Participants) | 2 | 2
  Erythrocytes 3, n=2,2 | 0 | 1
  Erythrocytes 7, n=2,2: number analyzed (Participants) | 2 | 2
  Erythrocytes 7, n=2,2 | 1 | 0
  Erythrocytes 9, n=2,2: number analyzed (Participants) | 2 | 2
  Erythrocytes 9, n=2,2 | 0 | 1
  Leukocytes 1, n=2,2: number analyzed (Participants) | 2 | 2
  Leukocytes 1, n=2,2 | 2 | 1
  Leukocytes 2, n=2,2: number analyzed (Participants) | 2 | 2
  Leukocytes 2, n=2,2 | 0 | 1

36. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Full 12-lead ECGs were recorded with the participant in a supine position. The number of participants with abnormal clinically significant ECG findings for worst case post-Baseline is presented.
Time Frame: Period 1: Up to Day 6; Period 2: Up to Day 10
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

37. Secondary Outcome: Number of Participants With Abnormal Spirometry Values
Description: Spirometry assessments were planned but not performed.
Time Frame: Period 1: Day -1; Period 2: Day 4
Population: Safety population.
Arm/Group | Nemiralisib 100 mcg | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Millimeter of mercury
  SBP | -1.2 (4.21)
  DBP | -0.5 (3.71)

39. Secondary Outcome: Change From Baseline in SBP and DBP When Single Inhaled Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose
Description: as for outcome 38
Time Frame: Baseline (Day 1, pre-dose) and Days 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Millimeter of mercury
  SBP, Day 2 | 0.2 (3.71)
  SBP, Day 4 | -1.2 (6.37)
  SBP, Day 6 | -2.6 (5.60)
  SBP, Day 8 | -1.8 (6.15)
  SBP, Day 10 | 1.4 (6.86)
  DBP, Day 2 | -1.0 (3.04)
  DBP, Day 4 | -0.7 (6.21)
  DBP, Day 6 | -3.5 (4.16)
  DBP, Day 8 | -3.4 (3.39)
  DBP, Day 10 | -0.5 (3.52)

40. Secondary Outcome: Change From Baseline in Pulse Rate When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered
Description: Pulse rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Beats per minute | -1.9 (8.83)

41. Secondary Outcome: Change From Baseline in Pulse Rate When Single Inhaled Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose
Description: as for outcome 40
Time Frame: Baseline (Day 1, pre-dose) and Days 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Beats per minute
  Day 2 | 1.9 (4.80)
  Day 4 | 3.2 (6.44)
  Day 6 | 1.4 (6.15)
  Day 8 | 3.5 (7.83)
  Day 10 | 2.3 (6.55)

42. Secondary Outcome: Change From Baseline in Respiratory Rate When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered
Description: Respiratory rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Breaths per minute | -0.4 (2.01)

43. Secondary Outcome: Change From Baseline in Respiratory Rate When Single Inhaled Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose
Description: as for outcome 42
Time Frame: Baseline (Day 1, pre-dose), Days 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Breaths per minute
  Day 2 | -1.3 (1.87)
  Day 4 | 0.3 (1.63)
  Day 6 | -0.5 (1.82)
  Day 8 | 0.1 (1.77)
  Day 10 | -0.5 (2.24)

44. Secondary Outcome: Change From Baseline in Temperature When Single Inhaled Oral Dose of Nemiralisib 100 mcg Administered
Description: Temperature of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Nemiralisib 100 mcg
Number analyzed (Participants) | 20
Celsius | 0.04 (0.188)

45. Secondary Outcome: Change From Baseline in Temperature When Single Inhaled Oral Dose of Nemiralisib 100 mcg Co-administered With Itraconazole 200 mg Repeated Dose
Description: as for outcome 44
Time Frame: Baseline (Day 1, pre-dose), Days 2, 4, 6, 8 and 10
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Itraconazole 200 mg and 100mcg Nemiralisib on Day 5
Number analyzed (Participants) | 20
Celsius
  Day 2 | -0.03 (0.205)
  Day 4 | -0.07 (0.239)
  Day 6 | -0.03 (0.266)
  Day 8 | -0.08 (0.234)
  Day 10 | -0.07 (0.213)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and adverse events (AEs) were collected up to Day 35
Description: AEs and SAEs were collected in the Safety Population.
Arm/Group | Nemiralisib 100 mcg | Nemiralisib 100 mcg With Itraconazole 200 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemiralisib 100 mcg (N=20) | Nemiralisib 100 mcg With Itraconazole 200 mg (N=20)
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03398421/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03398421/SAP_001.pdf